CLINICAL TRIAL: NCT06394128
Title: Study on the Curative Effect of Cangpo Liujun Prescription on Cancer-related Fatigue in Patients With Advanced Colorectal Cancer Undergoing Second-line Chemotherapy With Spleen Deficiency and Dampness Excess and Analysis of Intestinal Flora
Brief Title: Cangpo Liujun Prescription on Cancer-related Fatigue in Advanced Colorectal Cancer With Spleen Deficiency and Dampness Excess
Status: Recruiting | Phase: Phase 2 | Type: Interventional
Sponsor: First People's Hospital of Hangzhou (Other)
Responsible Party: Principal Investigator, Guokaibo, Dr., First People's Hospital of Hangzhou
Allocation: Randomized | Model: Parallel | Masking: Single | Purpose: Treatment
Other Study IDs: CPLJF
Record Dates: First submitted 2024-04-05; First posted 2024-05-01 (Actual); Last update posted 2024-05-01 (Actual); Status verified 2024-04

CONDITIONS: Cancer-Related Fatigue; Colorectal Cancer
MeSH Terms: conditions — Colorectal Neoplasms

STUDY DESIGN:
Who Masked: Participant
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

ARMS (2):
- Cangpo Liujun Prescription (Experimental): Cangpo Liujun Prescription composition: Rhizoma atractylodis 15g, Magnolia officinalis 12g, Tangerine peel 15g, Pinellia pinellia 12g, Codonopsis ginseng 15g, Rhizoma atractylodis macrocephalae 15g, Poria cocos 15g, Honey-fried licorice root 6g. It was taken during and between the treatments, in the morning and in the evening, 200ml each time, for 3 courses, and 1 course was 28 days.
  Interventions: Drug: Cangpo Liujun Prescription
- Placebo (Placebo Comparator): Cangpo Liujun Prescription granule mimics was made into a control placebo according to the content of 5% of the treatment group. It was taken during and between the treatments, in the morning and in the evening, 200ml each time, for 3 courses, and 1 course was 28 days.
  Interventions: Drug: Cangpo Liujun Prescription

INTERVENTIONS:
Drug: Cangpo Liujun Prescription — Based on the diagnostic criteria of spleen deficiency and dampness excess syndrome, Cangpo Liujun Prescription could be used to treat cancer-related fatigue in patients with advanced colorectal cancer undergoing second-line chemotherapy.
  Other Names: CPLJ

SUMMARY:
The goal of this clinical trial is to learn if Cangpo Liujun Prescription works to treat cancer-related fatigue in patients with advanced colorectal cancer undergoing second-line chemotherapy with spleen deficiency and dampness excess. It will also learn about the safety of Cangpo Liujun Prescription. The main questions it aims to answer are:

Does Cangpo Liujun Prescription improve the fatigue symptoms for participants? How about the relationship between taking Cangpo Liujun Prescription and distribution of intestinal flora?

Researchers will compare Cangpo Liujun Prescription to a placebo (a look-alike substance that contains no drug) to see if Cangpo Liujun decoction works to treat cancer-related fatigue in patients with advanced colorectal cancer undergoing second-line chemotherapy with spleen deficiency and dampness excess.

Participants will:

Take Cangpo Liujun Prescription or a placebo every day for 3 months Visit the clinic once every 2 weeks for checkups and tests Keep a diary of their symptoms Take blood samples to detect immune function and inflammatory factors Collected Feces for gut microbiota analysis

DETAILED DESCRIPTION:
1. Patients with advanced colorectal cancer undergoing chemotherapy constitute a significant demographic affected by cancer-related fatigue (CRF).

   CRF, as delineated by NCCN guidelines, is described as enduring, subjective physical, emotional, and/or cognitive weariness or fatigue related to cancer or its treatment, significantly interfering with daily life and function. It stands as one of the most common and severe accompanying symptoms among cancer patients, with durations extending up to five years for a quarter to a third of patients. The etiology of CRF is complex, with factors including tumor-related factors, treatment-related factors (surgery, radiotherapy, chemotherapy, immunotherapy, etc.), comorbidities (anemia, thyroid dysfunction, etc.), and psychosocial factors (anxiety, depression, etc.). CRF exerts various adverse effects on patients, significantly diminishing their quality of life, including changes in daily habits, decreased vitality, a sense of loss of control, social isolation, and exacerbation of other accompanying symptoms. Moreover, CRF may reduce patients' completion rates of anti-tumor treatment, consequently diminishing their survival periods, highlighting its substantial detrimental impact. Studies indicate that approximately 33% of colorectal cancer patients experience CRF after chemotherapy, with the incidence rising to two-thirds in advanced colorectal cancer patients, likely associated with multiple chemotherapy treatments and low nutritional status. Chemotherapy can lead to immunosuppression, tissue cell damage, and release of inflammatory cytokines. Among these, cytokines play a crucial role in CRF formation, inducing central fatigue through mechanisms such as anemia, cachexia, and disruption of the hypothalamic-pituitary-adrenal axis. Additionally, regimens such as oxaliplatin and its combinations (FOLFOX, FOLFIRI, FOLFOXIRI) used in colorectal cancer treatment can cause mitochondrial and energy homeostasis dysregulation, leading to skeletal muscle fatigue, with cumulative toxicity. Reduced energy intake due to chemotherapy often results in prolonged low nutritional status in colorectal cancer patients. Decreased synthesis of proteinaceous substances and accumulation of certain metabolites alter ATP metabolism within muscle cells, thereby precipitating peripheral fatigue.
2. The principal pathogenesis of cancer-related fatigue (CRF) in patients undergoing second-line treatment for colorectal cancer is spleen deficiency and dampness accumulation.

   Although ancient Chinese medical texts do not directly mention "colorectal cancer" or "tumors," traditional Chinese medicine has a deep-rooted understanding of similar symptoms associated with clinical manifestations, such as "intestinal tumors" and "accumulations," found in the "Inner Canon." The "Surgical Orthodoxies · Doctrine of Internal Infections" elucidates that spleen deficiency leads to the accumulation of damp toxins, which, over time, accumulate heat. This accumulation of damp-heat toxins flows into the intestines, resulting in poor local circulation of qi and blood and the coagulation of damp toxins into cancerous masses. Prolonged retention of tumors in the intestines depletes qi and injures body fluids, exacerbated by chemotherapy and targeted therapies, giving rise to a clinical presentation akin to traditional Chinese medicine's concept of "deficiency fatigue." This includes a series of symptoms such as visceral function decline, overall debilitation, weakness, lethargy, emaciation, and increased inclination toward sleep, aligning closely with the scope of CRF. The term "deficiency fatigue" was first documented by Zhang Zhongjing in "Synopsis of the Golden Chamber · Blood Stasis Deficiency Fatigue Disease Pulse Syndrome and Treatment," illustrating that spleen deficiency is the primary pathogenesis of deficiency fatigue and CRF. According to traditional Chinese medicine, CRF is predominantly characterized by deficiency patterns, often compounded with mixed patterns of deficiency and excess, with the affected organs primarily involving the spleen, lungs, liver, and kidneys, accompanied by pathological factors such as qi stagnation and damp turbidity. Second-line treatment patients with advanced colorectal cancer, following first-line chemotherapy or combined targeted therapy, often present with spleen and stomach deficiency, leading to inefficient transformation and transportation processes. The spleen has an inclination toward dryness while detesting dampness, yet internal damp evils originate and propagate due to the humid climate of the southern region, inducing internal dampness that exacerbates the deficiency of the spleen, resulting in a state of spleen deficiency and dampness accumulation within the body. This dampness, characterized by heaviness and turbidity, manifests as a sensation of head heaviness, overall lethargy, and heaviness and laziness in the limbs. Dampness, being a yin evil, easily obstructs the flow of qi and compromises yang qi, exacerbating spleen deficiency and intensifying the symptoms of deficiency fatigue. Hence, "spleen deficiency and dampness accumulation" constitute the primary pathogenesis of CRF in second-line treatment patients with colorectal cancer. The "Cangpo Liujun Prescription" is a commonly used prescription for the pattern of spleen deficiency and dampness accumulation, demonstrating certain efficacy in clinical prevention and treatment of CRF. Composed of Cang Zhu, Hou Po, Chen Pi, Ban Xia, Dang Shen, Bai Zhu, Fu Ling, and Gan Cao, this formula employs Cang Zhu and Hou Po to eliminate dampness and fortify the spleen, while Ban Xia and Chen Pi transform phlegm and regulate qi. Dang Shen, Bai Zhu, Fu Ling, and Gan Cao collectively tonify the spleen and boost qi, with all eight herbs synergistically promoting spleen health and dampness transformation, thereby ameliorating CRF-related symptoms. A preliminary retrospective study involving six patients with colorectal cancer who underwent first-line treatment and were planned for second-line treatment found that the Cangpo Liujun Prescription could reduce PFS-R scores, increase KPS scores, and improve patients' quality of life.
3. The differences in intestinal microbiota among colorectal cancer patients with different traditional Chinese medicine (TCM) patterns indicate that maintaining the stability of the microbiota is pivotal for alleviating cancer-related fatigue (CRF) symptoms.

   Research has increasingly shown the relationship between disruptions in the gut microbiota and various diseases. For instance, compared to healthy individuals, the abundance of Clostridium and Haemophilus genera is significantly higher in cases of Qi and Yin deficiency, while Bacteroides, Gemmiger, and Prevotella genera are more prevalent in patients with Phlegm-Dampness syndrome. Contrasting wet-heat syndrome with non-wet-heat syndrome individuals reveals a higher abundance of Veillonella, Coprococcus, and Acidaminococcus genera in the latter. Additionally, studies on a spleen deficiency rat model demonstrated that intervention with Si-Jun-Zi-Tang significantly improved symptoms such as eye squinting, hunched back, and lethargy, potentially by modulating the immune system and gut microbiota (mainly lactobacillus, Dorea, and Butyricimonas genera).

   Comparing late-stage colorectal cancer patients with early-stage ones, the former exhibit higher spleen deficiency scores, accompanied by a significant increase in Prevotella, Escherichia-Shigella, and Bacteroides genera, while the abundance of Clostridium sensu stricto is notably reduced. Furthermore, our team investigated the differences in intestinal microbiota between colorectal cancer patients with a deficiency of righteous Qi and those with an abundance of pathogenic factors. We found that, compared to the healthy control group, the abundance of Clostridium difficile was reduced in the deficiency of righteous Qi group, while lactobacillus abundance increased. In contrast, there was a decrease in Prevotellaceae abundance and a significant increase in Streptococcaceae in the group with an abundance of pathogenic factors, providing a biological basis for TCM syndrome differentiation and treatment in colorectal cancer.

   Current pharmacological treatments for CRF, such as psychostimulants (e.g., methylphenidate), modafinil, paroxetine, and dietary supplements (e.g., coenzyme Q10, L-carnitine, guarana), have not yet achieved satisfactory efficacy and are associated with certain side effects. With further research, it has been discovered that the composition of the intestinal microbiota is closely related to the severity of CRF. The central nervous system plays a crucial role in inducing CRF. Cancer cells disrupt the stability of the gut microbiota during their development, and gut microbiota imbalance can indirectly affect the central nervous system via the gut-brain axis, further exacerbating CRF. Inflammation may be the primary driving factor affecting the gut-brain axis. Therefore, maintaining the stability of the microbiota is crucial for alleviating CRF symptoms. Traditional Chinese medicine (TCM) and its active ingredients can regulate the composition of the gut microbiota, thereby influencing the reshaping of the tumor microenvironment in colorectal cancer treatment, and TCM has indeed been shown to significantly improve CRF-related symptoms, warranting further investigation.
4. Scientific hypothesis and research significance. Based on the preliminary research findings and literature review, our team posits a rational hypothesis: the administration of Cangpo Liujun Prescription (CPLJ) may ameliorate cancer-related fatigue (CRF) symptoms in advanced colorectal cancer patients with Spleen Deficiency and Dampness Excess (SDDE) type by rectifying chemotherapy-induced intestinal microbiota dysbiosis (IFI), thereby reducing the levels of inflammatory factors in the body and modulating the gut-brain axis (refer to Figure 1). We propose to include CRF patients with SDDE type late-stage colorectal cancer, randomly assigning them into two groups (CPLJ group and placebo group), and comparing differences in patients' Progression-Free Survival-Related (PFS-R) scores, traditional Chinese medicine syndrome scores, quality of life assessments, immune function tests, inflammatory factor assays, objective response rates (ORR), disease control rates (DCR), as well as intestinal microbiota, aiming to offer a novel effective approach for TCM treatment of CRF in late-stage colorectal cancer, to explore new biomarkers for CRF and its translational research, and to further enrich the microcosmic differentiation system of intestinal microbiota in SDDE type late-stage colorectal cancer patients.

ELIGIBILITY:
Inclusion Criteria:

(1) Diagnosis of stage IV colorectal cancer: confirmed by pathology or cytology; (2) Second-line treatment; (3) Clinical diagnosis of cancer-related fatigue; (4) Traditional Chinese medicine syndrome differentiation with spleen deficiency and damp excess; (5) PS score ≤2; (6) Age of 18-75 years old; (7) Predicted survival time ≥3 months; (8) Without other serious complications; (9) Non-pregnant and lactating patients; (10) Without allergic reaction to the ingredients in the prescription; (11) Agreed to participate in the study after informed consent, signed the informed consent form, and had good compliance.

Exclusion Criteria:

1) Conditions that may prevent the subjects from completing the clinical trial process, including but not limited to serious and difficult to control organic lesions or infection, heart failure, etc.; Patients with severe liver and kidney dysfunction (serum creatinine ≥1.5 times ULN; ALT or AST≥5 times ULN; Bilirubin ≥1.5 times ULN); (2) Combined with hematopoietic system diseases, such as anemia, requiring anemia correction drugs; (3) Receiving or preparing to receive treatment that may affect CRF; (4) Taking other drugs that may improve CRF; (5) Combined with tumors of other systems; (6) Mental illness or lack of independent behavior ability; (7) Cooperate with the investigators to complete the clinical investigation; (8) Pregnant, preparing to become pregnant or lactating women; (9) Participating in other clinical trials or have participated in other clinical trials within 3 months; (10) Alcohol and/or psychoactive substances, substance abusers and addicts; (11) According to the investigator's judgment, other lesions or conditions that may reduce or complicate the possibility of enrollment, such as frequent changes in work environment, unstable living environment, and other conditions that may cause loss to follow-up.

Ages: 18 Years to 75 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 48 (Estimated)
Dates: Start 2024-04-30 (Estimated); Primary Completion 2025-04-01 (Estimated); Study Completion 2026-04-01 (Estimated)

PRIMARY OUTCOMES:
The Revised Piper Fatigue Scale (PFS-R) | 3 months
  PFS-R included 22 items in total, which were divided into 4 dimensions: feeling, cognition, emotion and behavior. The behavioral dimension and cognitive dimension each contained 6 items, and the emotional dimension and feeling dimension each contained 5 items. Each item was scored on a scale of 0 to 10, and the total score was calculated by dividing the total score of all items by the number of items 22 to obtain the final score, with higher scores indicating more severe fatigue. The specific grading scale was 0-3 as mild, 4-6 as moderate, and 7-10 as severe. The severity of fatigue represented by each score was as follows: 0 indicated none, 1-3 mild, 4-6 moderate, and 7-10 severe.

SECONDARY OUTCOMES:
Traditional Chinesne medicine syndrome score | 3 months
  According to the criteria of cancer-related fatigue of spleen deficiency and damp excess type, the clinical symptoms and signs of the patients were observed, including fatigue, less qi and lazy speech, nausea and lethargy, numbness in the chest cavity, dull abdominal pain, difficulty in relieving or loose stool, spitting wet phlegm, distension after eating, light mouth without thirst, heavy head and body, light fat tongue, white or thin white mossy, thin or slippery pulse.The Traditional Chinesne medicine syndrome scores represented by each score were as follows: 0 for none, 1-3 for mild, 4-6 for moderate, and 7-10 for severe.
Assessment of quality of life | 3 months
  The quality of life was evaluated according to the Karnofsky performance status scale (KPS) standard. Including 0-100 points, Karnofsky score above 80 points is generally considered to be independent, that is, self-care level. 50-70 was divided into semi-independent, that is, semi-independent life. A score below 50 is dependent, meaning you need help in your life.
Immune function tests | 3 months
  Peripheral blood was collected from the patients, and the percentage and absolute count of lymphocyte subsets (CD3+T cells, CD4+T cells, CD8+T cells, NK cells and B cells) were detected by flow cytometry to evaluate the immune function.
Detection of inflammatory factors | 3 months
  The levels of interleukin (IL) -1β, IL-6, interferon (IFN) and tumor necrosis factor-α (Tnf-α) in peripheral blood were detected by enzyme-linked immunosorbent assay (ELISA).
Objective Response rate (ORR) and disease control rate (DCR) | 3 months
  According to Response Evaluation Criteria in Solid Tumors (RECIST), the objective effect of tumor relief was evaluated and divided into complete relieve (CR), partial relieve (PR) and stable disease (stable disease). SD), progress disease (PD), ORR (%) = (CR+PR)/total cases ×100%. DCR (%) = (CR+PR+SD)/total cases ×100%.
Detection of gut microbiota | 3 months
  Stool samples were collected from 48 patients before and after medication for 16S rDNA sequencing, and sequence clustering was performed using VSEARCH
Toxic and side effect (Blood routine) | 3 months
  The level of bone marrow suppression can be divided into grade 0-IV according to WHO. Grade 0 : white blood cell count greater than or equal to 4.0×10^9 /L, hemoglobin concentration greater than or equal to 110g/L, platelet greater than or equal to 100×10^9 /L. Grade Ⅰ : white blood cell count (3.0-3.9)×10^9 /L, hemoglobin concentration 95-100 g/L, platelet count (75-99)×10^9 /L. Grade Ⅱ : white blood cell count (2.0-2.9)×10^9 /L, hemoglobin concentration 80-94 g/L, platelet count (50-74)×10^9 /L. Grade Ⅲ : white blood cell count (1.0-1.9)×10^9 /L, hemoglobin concentration 65-79g/L, platelet (25-49)×10^9 /L. Grade Ⅳ : white blood cell count (0-1.0)×10^9 /L, hemoglobin concentration <65g/L, platelet <25×10^9 /L.
Toxic and side effect (liver function) | 3 months
  Child-Pugh classification of liver function, known as Child-Pugh classification, is A commonly used index to evaluate liver reserve function in patients with cirrhosis. It is mainly divided into grade A, B and C according to a variety of indicators by scoring method. The main indicators included serum bilirubin, serum albumin, prothrombin time, and whether complicated with ascites and hepatic encephalopathy. According to the level of increase or decrease in the index, as well as the degree of severity of complications, you can add 1 point, 2 points or 3 points respectively, usually the higher the total score, the worse the liver reserve function.
Toxic and side effect (kidney function) | 3 months
  kidney function is divided into 1-5 stages according to the degree of renal function damage and glomerular filtration rate. Stage 1: the performance of renal function is basically normal, and the glomerular filtration rate is 90-120 ml /min. Stage 2: At this time, the patient may have mild renal impairment, with a decreased glomerular filtration rate, between 60 and 89mL/min. Stage 3: Renal function has been significantly impaired, and the glomerular filtration rate can drop to 30 to 59mL/min. For patients with chronic kidney disease, stage 3a glomerular filtration rate is 45 to 59mL/min. 3b 30-44ml/min, without timely intervention, may progress rapidly to renal failure stage. Stage 4: At this time, the patient's renal function has severely declined, and the glomerular filtration rate is only 15-29 ml /min. Stage 5: enter the end-stage renal disease, glomerular filtration rate < 15mL/min, most patients need dialysis maintenance.

CONTACTS AND LOCATIONS:
Locations (1):
- Hangzhou First People' Hospital, Hangzhou, Zhejiang, China

IPD SHARING:
Plan to Share IPD: No